CLINICAL TRIAL: NCT02350842
Title: Triple-site Biventricular Stimulation in the Optimization of Cardiac Resynchronization Therapy (CRT)
Brief Title: Triple-site Biventricular Stimulation in the Optimization of CRT
Acronym: TRIUMPH-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICSY02
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
Keywords: non-Left Bundle Branch Block morphology; Triple-site biventricular pacing; cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple-site biventricular pacing (Experimental): Triple-site biventricular pacing with individual optimization of the placement of the third lead by peri-operative echo guidance. Devices used will be the Sorin, locally approved and commercially available Paradym SonR Tri-V CRT-D.
  Interventions: Device: triple-site biventricular pacing with peri-operative echo guidance
- Standard biventricular pacing (Active Comparator): Standard biventricular pacing (1RV/1LV) through classical implantation procedure without peri-operative optimization. Devices used will be locally approved and commercially available Sorin implantable cardioverter defibrillators.
  Interventions: Device: standard biventricular pacing

INTERVENTIONS:
Device: triple-site biventricular pacing with peri-operative echo guidance — placement of the third lead by peri-operative echo guidance.
  Arms: Triple-site biventricular pacing
Device: standard biventricular pacing — standard biventricular pacing without optimization by echo guidance
  Arms: Standard biventricular pacing

SUMMARY:
Cardiac resynchronization is a recommended therapy for patients with advanced heart failure, under optimized medical treatment with reduced left ventricular ejection fraction and prolonged QRS, nevertheless, still 30% of the population do not respond to standard biventricular implantation.

Non-response can be explained by a combination of factors including sub-optimal patient selection, placement of the pacing lead over a zone of slow conduction, insufficient correction of mechanical dyssynchrony including sub-optimal lead implantation. Few data distinguish true non-responders from patients in which effective resynchronization was not delivered through standard biventricular implantation.

Triple-site cardiac resynchronization pacing (stimulation at three ventricular sites) has been proposed to improve synchrony and thus the response rate in (Cardiac Resynchronisation Therapy) CRT recipients.

DETAILED DESCRIPTION:
The frequent failure of CRT in non-Left Bundle Branch Block (non-LBBB) patients is suspected to be due to more complex and heterogeneous forms of electrical/mechanical dyssynchronies needing more complex and individualized pacing configurations to be corrected.

Acute studies during implant show that standard biventricular pacing provides optimal mechanical improvement only in a minority of patients. In a peri-operative echo-guided leads placement procedure most of non-improved patients could be successfully mechanically resynchronized. A significant number of patients required optimized placement of right ventricular (RV) lead and/or triple-site configurations.

These studies led to the hypothesis that more complex and individualized pacing configurations (Triple-site biventricular) might increase the number of responders to CRT.

To assess this hypothesis, this study will be conducted in Class II-ambulatory IV patients indicated for CRT with wide QRS (≥ 140 ms) and non-LBBB. Patients will be randomized in a 1:1 configuration:

* Standard biventricular pacing (1 right ventricular/1 left ventricular (1RV/1LV)) through classical implantation procedure without peri-operative optimization
* Triple-site biventricular pacing with individual optimization of the placement of the third lead by peri-operative echo guidance.

The objective of the optimization process is to improve LV efficiency and to decrease the left pre-ejection interval (LPEI, defined as the time interval between the onset of QRS and the onset of LV ejection) as much as possible compared with a standard biventricular configuration by moving a second right ventricular lead at different locations.

LPEI is simple to measure, with good inter- and intra-observer reproducibility and its utility has previously been strongly suggested.

Reduction in LPEI results in decreased duration of ventricular systole and is associated with improved LV filling and reduced interventricular delay.

The primary objective of this study is to demonstrate that individually optimized, triple-site biventricular pacing is superior to standard biventricular pacing in reverse ventricular modeling as demonstrated by Echo Left Ventricle End-Systolic Volume (LVESV) at 1 year in patients with non-LBBB morphology without increasing the risk of serious procedure and/or device related adverse events at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Stable heart failure with New York Heart Association (NYHA) functional class II, III or ambulatory IV
* Stable optimized medical regimen according to medical guidelines (No change in heart failure medication for at least 1 month prior to enrollment)
* Left ventricular ejection fraction (LVEF) ≤ 35%
* Intrinsic QRS duration ≥ 140 msec
* Non-typical left bundle branch block (LBBB) morphology on 12-lead surface ECG
* Signed and dated informed consent

Exclusion Criteria:

* Typical LBBB according to Strauss criteria
* Unstable heart failure
* Permanent or long-lasting persistent Atrial Fibrillation
* Unstable angina, acute Myocardial Infarction (MI), Coronary Artery Bypass-Grafting (CABG), or Percutaneous Transluminal Coronary Angioplasty (PTCA) within 90 days prior to enrollment (intervention)
* Conventional pacemaker indication
* Previous implant with a pacemaker or an Implantable Cardioverter-Defibrillator (ICD)
* Renal Failure (Glomerular filtration rate (GFR) < 30 ml/min/1.73m2)
* Pregnant women
* Already included in another clinical study that could confound the results of this study
* Life expectancy < 12 months
* Mechanical heart valve or indication for valve repair or replacement
* Recent Cerebro-Vascular Accident (CVA) or Transient Ischemic Attack (TIA) (within the previous 3 months)
* Heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
TriV pacing is superior to standard BiV pacing in reversing ventricular modeling as demonstrated by Echo LVESV at 12 months in pts. with non LBBB without increasing the risk of serious events at 30 days. | 12 months
  The efficacy endpoint for this study is the change in LVESV at twelve months post-implant between individually optimized, triple-site biventricular pacing and standard biventricular pacing.
  LVESV is a standard marker of CRT effectiveness1. Echocardiographic data collected at twelve months follow-up will document the evolution of LVESV as compared to baseline in order to assess reverse ventricular remodeling.
  The safety endpoint for this study is the rate of all serious procedure and/or device related events reported at thirty days post-implant.

SECONDARY OUTCOMES:
Evaluate serious device related complications at six and twelve months post-procedure. | 6 and 12 months
  A safety assessment will be performed, including all reported events collected for all enrolled patients.
Evaluate reverse ventricular remodeling response based on additional echocardiographic measures | 6 and 12 months
  Change in LV volumes and LV ejection fraction will be evaluated as part of reverse remodeling response, based on echocardiographic measurements:
  * LVESV at 6 months
  * LVEDV at 6 and 12 months
  * LVEF at 6 and 12 months
Evaluate patient's clinical status considering New York Heart Association (NYHA) functional class improvement | 6 and 12 months
  A patient's clinical status will be evaluated considering:
  * NYHA functional class improvement - The evaluation of the NYHA classification consists of reporting the percentage of patients who improved at least one NYHA class at each follow-up post-implant.
  * Death from any cause - The reporting of deaths occurred consists of the percentage of dead patients, the causes of death, the time to death and survival curves.
  * HF-related hospitalizations, as defined in section 15.4.
  * The incidence of serious device related events assessed at six and twelve months.
Evaluate mortality and serious heart failure (HF) events during the procedure through discharge and at the different follow-up time-points. | 1, 6 and 12 months
  A safety assessment will be performed, including all reported events collected for all enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Daubert, MD, Principal Investigator — Hôpital Pontchaillou-CHU Rennes, France
Locations (14):
- France (8):
  - CHRU Hopital Sud, Amiens
  - Clinique Rhone Durance, Avignon
  - Hopital Jean Minjoz Besançon, Besançon
  - CHRU Brest, Brest
  - Groupe hospitalier Paris Saint-Joseph, Paris
  - CHU Poitiers, Poitiers
  - CHU Hôpital Charles Nicolle, Rouen
  - CHU Toulouse, Hopital Rangueil, Toulouse
- Universitaetsklinikum Schleswig Holstein, Kiel, Germany
- Humanitas Cliniche Gavazzeni spa, Bergamo, Italy
- Isala Zwolle, Zwolle, Netherlands
- CHCL - Hospital Santa Marta, Lisbon, Portugal
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario La Fe, Valencia